CLINICAL TRIAL: NCT05056389
Title: Normothermic Intraperitoneal Chemotherapy - Long Term in Peritoneal Metastases From Colorectal Cancer - Feasibility Study (NIPEC-OXA)
Brief Title: Normothermic Intraperitoneal Chemotherapy - Long Term in Peritoneal Metastases From Colorectal Cancer (NIPEC-OXA)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Mariusz Goscinski, Principal Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202644
Record Dates: First submitted 2021-09-09; First posted 2021-09-24 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Peritoneal Metastases; Colo-rectal Cancer
Keywords: NIPEC-LT; Oxaliplatin; CRS; HIPEC
MeSH Terms: conditions — Colonic Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Feasibility study with 20 eligible patients with peritoneal metastases from colorectal cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NIPEX-OXA arm (Experimental): 20 patients treated with NIPEC-OXA after CRS and HIPEC.
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — Administration of oxaliplatin intraperitoneally
  Other Names: Intraperitoneal catheter

SUMMARY:
Feasibility study regarding 20 Patients with peritoneal metastases from colorectal cancer treated with cytoreductive surgery and HIPEC and subsequently with 4 courses of normothermic intraperitoneal chemotherapy - long term (NIPEC-OXA) with oxaliplatin.

DETAILED DESCRIPTION:
Primary endpoint: to determine if the administration of additional i.p. chemotherapy for a period of 9 weeks after completed CRS and HIPEC is a safe procedure to be used in the future in a formal randomised trial. The toxicity of the chemotherapy given through i.p. during NIPEC-OXA courses will be analysed throughout the entire treatment period and a subsequent 3-month follow-up period.

Secondary endpoints:

1. Intra-abdominal chemotherapy drug distribution 7-14 days after CRS and HIPEC and before the 4th NIPEC-OXA course
2. Surgical complications after CRS, HIPEC and NIPEC-OXA until 3 months after the last NIPEC-OXA course
3. Disease-free survival (DFS)
4. Overall survival (OS)

Exploratory endpoint: quality of life

Estimated date of first patient enrolled: 3rd quarter of 2021 Anticipated recruitment period: 1,5 years Estimated treatment completion date of last patient: 1st quarter of 2023 Expected treatment duration per patient: 9 weeks Expected follow-up period per patient: 3 months after the last NIPEC-OXA procedure

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years
* Able to provide written, informed consent regarding expected cooperation during treatment and follow-up according to ICH GCP, and national/local regulations
* Histologically verified CRC
* Histologically verified and/or radiologically/clinically suspected PM from CRC
* Synchronous or metachronous PM from CRS

  * If neoadjuvant oxaliplatin-containing chemotherapy is administrated, patients with absence of progressive disease (assessed by CT)
  * In metachronous cases: if adjuvant oxaliplatin-containing chemotherapy, the interval between oxaliplatin- containing adjuvant chemotherapy and diagnosis of PM must be >6 months
* Intraperitoneal tumour burden amenable to CRC and HIPEC with Peritoneal Cancer Index (PCI40) ≤ 20, assessed at the time of surgery
* Absence of other metastatic sites, i.e. liver, lungs, central lymph nodes
* Completeness of Cytoreduction (CC) score of 0 is required
* Eastern Cooperative Oncology Group (ECOG) Performance Status either 0 or 141
* Women of childbearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, should have a negative urine- or serum pregnancy test within 72 hours prior to receiving the 1st dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* WOCBP should be willing to use 1 highly effective method of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.
* Men in a sexual relationship with a WOCBP must agree to use a condom starting with the 1st dose of study therapy through 120 days after the last dose of study therapy. In case of female partner of child-bearing potential, the female partner should use 1 highly effective contraception method as defined in section 5.1.5 - "Other considerations".

Exclusion Criteria:

* Has a history of hypersensitivity to oxaliplatin or to any of the excipients listed in the SmPC section 6.1
* Has myelosuppression before starting treatment, ie number of neutrophils granulocytes <1.0 x 109/l and/or number of platelets <75 x 109/l
* Has peripheral sensitive neuropathy with functional outcomes before starting treatment
* Has severe renal impairment (creatinine clearance < 30 ml min) (see the SmPC section 5.2).
* Concurrent or previous diagnosis of invasive cancer within 5 years
* Psychiatric or addictive disorder or other medical condition that would preclude the patient from meeting the trial requirements
* Participation in another cancer clinical trial
* Patients who, according to current guidelines will be offered i.v. adjuvant therapy
* Significant cardiac or other medical illness that would limit activity or survival, such as severe congestive heart failure, unstable angina, or serious cardiac arrhythmia
* Alcohol or drug abuse
* Any reason why, in the opinion of the investigator, the patient should not participate
* Has a known history of Human Immunodeficiency Virus (HIV)
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected)
* Is pregnant or breastfeeding, or expecting to conceive or father children within the project duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events after Intraperitoneal Chemotherapy Administration (NIPEC-OXA) | Throughout the entire treatment period, including a 3-month follow-up
  Common Terminology Criteria for Adverse Events v. 5
Number of Participants with Surgical Complications after CRS, HIPEC and NIPEC-OXA | Throughout the entire treatment period, including a 3-month follow-up
  Clavien-Dindo classification

SECONDARY OUTCOMES:
Number of Participants with Optimal, Suboptimal and Missing Fluid Distribution in the Abdomen Injected Through 2 I.P. Catheters | 7-14 days after CRS and HIPEC and before the 4th NIPEC-OXA course
  CT scans with intraperitoneal contrast

CONTACTS AND LOCATIONS:
Overall Officials: Mariusz Goscinski, MD.PhD., Principal Investigator — Oslo University Hospital, The Norwegian Radium Hospital
Locations (1):
- The Norwegian, Radium Hospital, Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
The sponsor's representatives (e.g. monitors, auditors) and/or regulatory authorities will be allowed access to source data for source data verification in which case a review of those parts of the hospital records relevant to the study may be required.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data of the study will be kept 15 years after the end of the study according Norwegian law.
Access Criteria: Access to the data has to be approved by the PI.